CLINICAL TRIAL: NCT07038525
Title: A Non-Inferiority Randomized Controlled Trial Comparing the Effectiveness of Online Versus In-Person Suturing Training Among Medical Students in a Low Resource Setting
Brief Title: Online vs. In-Person Suturing Training: A Non-Inferiority Randomized Controlled Trial in a Low-Resource Setting
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diala Burjak (Other)
Responsible Party: Sponsor-Investigator, Diala Burjak, MD, Yarmouk University
Organization: Yarmouk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LYD-RCT001
Record Dates: First submitted 2025-05-16; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Suture Techniques; Training Effectiveness; Online Education; Student Education; Hands-on Training
Keywords: suturing skills; surgical education; online medical training; hands-on workshop; medical student; simulation-based learning; OSATS; low-resource setting; RCT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In person suturing training (Experimental): Participants in this arm will attend a live, instructor-led suturing training session using standardized kits. The session will involve hands-on practice under direct supervision. The curriculum and assessment criteria are consistent with the online arm to ensure parity in instructional content.
  Interventions: Other: Suturing training
- Online suturing training (Experimental): Participants in this arm will receive access to a pre-recorded instructional video and practice independently using identical kits. After completing the training, participants will receive real-time feedback via Zoom from a trainer. Instructional content and assessment tools are standardized across both groups.
  Interventions: Other: Suturing training

INTERVENTIONS:
Other: Suturing training — This intervention involves basic suturing skills training delivered either in-person or online. In the in-person group, participants receive live instruction and hands-on supervision. In the online group, participants watch a standardized video tutorial and receive remote feedback via Zoom. All participants use identical suturing kits and are evaluated using the same OSATS checklist by a blinded assessor. The content and learning objectives are standardized across both formats.
  Other Names: Suturing skills workshop

SUMMARY:
The goal of this clinical trial is to assess whether online suturing training is non-inferior to in-person training in developing suturing skills among medical students at Yarmouk University in a low-resource setting.

The main questions it aims to answer are:

* Is online suturing training as effective as in-person training in developing practical skills (as measured by OSATS scores)?
* Does online training result in comparable knowledge improvement compared to in-person training (as measured by MCQ scores)?

Researchers will compare the online video-based training with Zoom feedback to live instructor-led in-person training to see if the online approach is not clinically inferior in terms of skills and knowledge acquisition.

Participants will:

* Complete pre-assessment and informed consent
* Be randomly assigned to one of the two training groups using stratified block randomization
* Participate in a suturing workshop either in-person or via online video and Zoom feedback
* Complete a post-assessment including OSATS-evaluated performance and MCQ test

Allocation concealment will be maintained, and the OSATS scores will be assessed by a blinded evaluator using a standardized checklist.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effectiveness of online versus in-person suturing training among medical students in a low-resource setting. Suturing is a core skill expected of medical students and a critical component of surgical training. With increasing demand for flexible and accessible medical education, online learning platforms have gained popularity. However, the comparative effectiveness of virtual training versus traditional in-person instruction in delivering procedural skills remains underexplored, particularly in low-resource environments.

This trial is designed as a phase II, parallel-group, non-inferiority randomized controlled trial with stratified block randomization and blinded outcome assessment. The goal is to determine whether online video-based suturing instruction, supplemented with real-time feedback via Zoom, is non-inferior to traditional in-person training in achieving technical skill acquisition, as measured by the Objective Structured Assessment of Technical Skills (OSATS).

Study participants are pre-clinical and clinical medical students from Yarmouk University who voluntarily consent to participate and complete all phases of the study. Participants will be stratified based on prior suturing experience (Yes/No) and randomly assigned in blocks of 4 or 6 to ensure balanced distribution across both training arms.

Allocation concealment is preserved through a standardized process: participants provide informed consent and complete baseline assessments before group assignment is revealed. The intervention is delivered in one of two formats, with both groups using identical suturing kits and standardized instructional material to reduce variability.

The in-person group receives live instructor-led training during a hands-on session.

The online group receives a pre-recorded instructional video and practices independently using the kit, followed by live Zoom-based feedback from a trainer.

Following the intervention, all participants are assessed via two primary methods:

* OSATS checklist, completed by a blinded evaluator based on video recordings of each participant's performance.
* Knowledge assessment, consisting of a five-question multiple choice test administered before and after the training to measure knowledge gain.

The OSATS tool used is a standardized and validated checklist evaluating multiple technical domains such as instrument handling, suture technique, and tissue approximation. The total OSATS score, which ranges based on the number of checklist items scored on a 1-5 scale, serves as the primary outcome. Knowledge scores (0-5) serve as the secondary outcome.

Statistical analysis will follow a pre-specified non-inferiority framework. Normality of score distributions will be assessed using Shapiro-Wilk tests. If assumptions are met, independent t-tests and 95% confidence intervals will be used to assess non-inferiority; if not, non-parametric alternatives (e.g., Mann-Whitney U tests) will be used. Sensitivity analyses will confirm robustness of findings using both parametric and non-parametric approaches. Within-group changes in knowledge scores will be analyzed using paired t-tests or Wilcoxon signed-rank tests, as appropriate.

To reduce potential bias, evaluator blinding is strictly maintained and only one evaluator is used to eliminate inter-rater variability. The use of standardized materials, identical kits, and consistent checklists across both groups ensures fairness and fidelity to protocol.

This study will serve as a pilot non-inferiority trial, intended to generate effect size estimates and assess the feasibility of larger-scale implementation in similar low-resource environments. While the planned sample size of 48 participants (24 per arm) may not detect moderate effect sizes with high power, it is sufficient to detect large differences and inform the design of future trials.

The broader educational aim of this trial is to provide insight into how surgical education can be adapted to virtual or remote learning formats without compromising quality, especially in regions where traditional instruction is limited by geographic, financial, or institutional constraints. Results may inform both local and international medical education strategies and support the development of cost-effective, scalable solutions to procedural training.

This project is conducted under the Live Your Dream (LYD) educational initiative and is fully self-funded by the investigator. No external funding or institutional sponsorship has been obtained. Results will be disseminated through academic conferences and peer-reviewed publication.

ELIGIBILITY:
Inclusion Criteria:

* Medical students (Yarmouk university)
* Signed informed consent

Exclusion Criteria:

* Incomplete workshop attendance
* Technical issues that hinder full participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
Total OSATS Score (Objective Structured Assessment of Technical Skills) | Within 2 days post-intervention
  The OSATS score will assess practical suturing skills using a standardized checklist across multiple domains (e.g., instrument handling, suture technique, knot tying). Each item is scored on a 1-5 ordinal scale, and scores are summed to create a total OSATS score. The evaluation will be conducted by a blinded assessor based on video recordings. The total score will be treated as a continuous variable if normality is satisfied and will serve as the primary outcome in assessing non-inferiority between the online and in-person training groups.

SECONDARY OUTCOMES:
Knowledge Assessment Score (Pre/Post MCQ) | Immediately before and after intervention (3 days total)
  Participants will complete a five-question multiple choice test before and after the suturing training. Each question is scored as correct (1) or incorrect (0), with a total score ranging from 0 to 5. This outcome evaluates knowledge acquisition related to suturing principles and techniques. Group differences in post-test scores, as well as within-group pre-post improvement, will be analyzed using appropriate statistical tests based on distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Diala Burjak, MD, Principal Investigator — NYC Health + Hospitals/ Elmhurst Hospital
Locations (1):
- Jordan Medical Association, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that will be shared include OSATS scores, pre- and post-intervention knowledge assessment scores, and basic demographic information (age, gender, clinical year, prior suturing experience). Data will be shared for academic research purposes upon reasonable request following publication of the main results. No personally identifiable information will be included. Access requests should be submitted to the Principal Investigator via email.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting documents (study protocol and informed consent form) will be made available within 6 months after publication of the primary results. Data will remain available for at least 3 years following release, or longer upon request.
Access Criteria: Qualified researchers, academic institutions, or organizations conducting health education or surgical training research may request access to the IPD and supporting documentation. Requests should include a research proposal and intended use. Data will be shared in de-identified format upon approval by the Principal Investigator and may be transmitted via secure email or file-sharing platforms.